CLINICAL TRIAL: NCT00580671
Title: Behavioral Treatment of Adolescent Marijuana Use
Brief Title: Treatment for Adolescent Marijuana Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Alan J. Budney, Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 75185; 5R01DA015186-07 (NIH); 5R01DA015186-08 (NIH)
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Results first posted 2013-06-05 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-07

CONDITIONS: Marijuana Abuse
Keywords: Adolescent Marijuana Abuse
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MET/CBT+CM/BPT (Experimental): Integrated psychosocial counseling. 14 weekly session. Twice weekly urine testing. Abstinence-based incentives based on urine test results. 14 weekly behavioral parenting sessions.
  Interventions: Behavioral: MET/CBT; Behavioral: CM; Behavioral: BPT
- MET/CBT+CM (Experimental): Integrated psychosocial counseling. 14 weekly sessions. Twice weekly urine testing. Abstinence-based incentives based on urine test results.
  Interventions: Behavioral: MET/CBT; Behavioral: CM
- MET/CBT (Active Comparator): Integrated psychosocial counseling. 14 weekly sessions.
  Interventions: Behavioral: MET/CBT

INTERVENTIONS:
Behavioral: MET/CBT — Weekly Individual Counseling Sessions
Behavioral: CM — Abstinence-based incentives delivered contingent on drug-negative urine test results.
  Arms: MET/CBT+CM; MET/CBT+CM/BPT
Behavioral: BPT — Behavioral parent training involve 14 weekly counseling curriculum to improve parenting skills.
  Arms: MET/CBT+CM/BPT

SUMMARY:
Marijuana remains the most prevalent illicit substance used by adolescents and the number of adolescents receiving treatment for marijuana abuse more than tripled during the last decade. A small number of clinical trials suggest that family-based and individual interventions have efficacy for treating adolescent substance abuse. However, even with these interventions most adolescents fail to reduce their substance use substantially, thus, there remains much room for improvement of treatment services. The overarching goal of this project is to develop and test novel behavioral treatments to enhance treatment outcome in this important treatment population, and in so doing, learn more about mechanisms of change that have broader implications for addiction science. In our initial Stage IB project "Behavioral Treatment for Adolescent Marijuana Abuse", we created, manualized, and pilot tested a unique contingency-management (CM) intervention that combined abstinence-based voucher incentives with contingency management training for parents. A small randomized, clinical trial provided encouraging results. When added to a commonly used cognitive-behavior therapy, CM improved rates of sustained abstinence during treatment. Adolescents receiving this intervention were less likely to relapse over the 9-month follow-up period, however this finding was not as robust as the observed during treatment effects, most likely due to the small sample size and associated low power to detect effects. Despite strong indicators of the efficacy of this CM intervention, there remained room for improvement in increasing rates of treatment response and reducing rates of relapse. Hypothesized mediators and moderators of change indicated that changes in parenting had direct effects on post-treatment marijuana abstinence outcomes, and that abstinence early in treatment was a robust predictor of the CM treatment effect. This proposal will systematically replicate and extend these findings. A Stage II trial will compare three treatment conditions: (1) cognitive behavior therapy (CBT only); (2) CBT plus CM; and (3) CBT plus an enhanced CM model targeting increased early abstinence rates, parenting skills, and maintenance of effects. Replicating the initial demonstration of the positive effects of CM will extend the scientific evidence for use of CM to increase treatment efficacy for substance-abusing adolescents. Testing an enhanced CM model will determine if modifications that are consistent with the underlying behavioral principles and empiricism supporting CM interventions can result in improved outcomes. Last, assessment of potential mechanisms of action, particularly parenting, adolescent psychopathology and impulsivity, will provide scientific information directly relevant to future development of more effective intervention and prevention models of adolescent substance abuse, and will inform us about fundamental mechanisms operating in drug-dependence.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 18 years old (if 18, they must attend high school and live at home)
* Report using marijuana during the previous 30 days or provide a marijuana- positive urine test
* Meet criteria for cannabis abuse or dependence
* Have a parent/guardian who can participate
* Live within a 30-minute driving range from the clinic

Exclusion Criteria:

* Currently meet DSM criteria for dependence on alcohol or other illicit drugs other than marijuana (use/abuse of other drugs will not be excluded)
* Exhibit active psychosis
* Have severe medical or psychiatric illness limiting participation
* Are pregnant or breast-feeding (youth only)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 153 (Actual)
Dates: Start 2007-11; Primary Completion 2012-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Budney, Ph.D., Principal Investigator — Dartmouth College
Locations (1):
- Geisel School of Medicine at Dartmouth, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] Kamon J, Budney A, Stanger C. A contingency management intervention for adolescent marijuana abuse and conduct problems. J Am Acad Child Adolesc Psychiatry. 2005 Jun;44(6):513-21. doi: 10.1097/01.chi.0000159949.82759.64. PMID 15908833
- [Derived] Stanger C, Ryan SR, Scherer EA, Norton GE, Budney AJ. Clinic- and home-based contingency management plus parent training for adolescent cannabis use disorders. J Am Acad Child Adolesc Psychiatry. 2015 Jun;54(6):445-53.e2. doi: 10.1016/j.jaac.2015.02.009. Epub 2015 Feb 28. PMID 26004659

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment opened in November 2007 and closed in February 2011. Participants were referred to the study for substance abuse treatment by school administrators, the juvenile justice system, community therapists, physicians or were self-referred. The study took place at an outpatient psychiatry clinic.
Pre-assignment Details: Clients were enrolled into the study and assessed for eligibility, if eligible they were given the choice to proceed. Reasons for ineligibility included no marijuana (MJ) use in past 30 days, failure to meet MJ abuse/dependence criteria, met dependence for another substance, no parent participant, plans to move away, low IQ
Groups:
- MET/CBT+CM/BPT: Motivational Enhancement Therapy (MET)/ Cognitive Behavior Therapy (CBT) + Contingency Management (CM) / Behavioral Parent Training (BPT)
- MET/CBT+CM: Motivational Enhancement Therapy (MET)/CBT+CM
- MET/CBT: Motivational Enhancement Therapy (MET)/CBT
Period: Overall Study
Arm/Group | MET/CBT+CM/BPT | MET/CBT+CM | MET/CBT
Started | 51 | 51 | 51
Completed | 35 | 35 | 34
Not Completed | 16 | 16 | 17

BASELINE CHARACTERISTICS:
Groups:
- MET/CBT+CM/BPT: Motivational Enhancement Therapy (MET)/CBT+CM/BPT
- Total: Total of all reporting groups
Arm/Group | MET/CBT+CM/BPT | MET/CBT+CM | MET/CBT | Total
Number analyzed (Participants) | 51 | 51 | 51 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 51 | 51 | 51 | 153
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (1.4) | 15.9 (1.3) | 15.7 (1.3) | 15.8 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 4 | 17
  Male | 44 | 45 | 47 | 136
Region of Enrollment [Number; unit: participants]
  United States | 51 | 51 | 51 | 153

OUTCOME MEASURES:

1. Primary Outcome: Marijuana Abstinence (2 Weeks or Greater)
Description: Percentage of participants who achieved 2 continuous weeks of marijuana abstinence as verified by twice weekly urine testing during the 14 weeks of treatment.
Time Frame: Testing done twice weekly for 14 weeks.
Measure: Number; unit: percentage of participants
Arm/Group | MET/CBT+CM/BPT | MET/CBT+CM | MET/CBT
Number analyzed (Participants) | 51 | 51 | 51
percentage of participants | 72.5 | 68.6 | 45.1

2. Secondary Outcome: Proportion of Days of Marijuana Abstinence Across All Days of Treatment (14 Weeks)
Description: This reflects the mean proportion of days of marijuana abstinence for each participant
Time Frame: This is for the proportion of days abstinent across the entire 14-week treatment period. Self-report data are collected twice weekly during treatment to obtain a cumulative proportion
Population: Those participants with data on at least 80 days of the 91 days of treatment were used in this analysis.
Measure: Mean (Standard Deviation); unit: proportion of marijuana abstinent days
Arm/Group | MET/CBT+CM/BPT | MET/CBT+CM | MET/CBT
Number analyzed (Participants) | 49 | 44 | 45
proportion of marijuana abstinent days | .8058 (.29419) | .8162 (.29143) | .7915 (.26115)

3. Primary Outcome: Marijuana Abstinence (4 Weeks or Greater)
Description: Percentage of participants who achieved 4 continuous weeks of marijuana abstinence as verified by twice weekly urine testing during the 14 weeks of treatment.
Time Frame: Twice weekly urine tests for 14 weeks.
Measure: Number; unit: percentage of participants
Arm/Group | MET/CBT+CM/BPT | MET/CBT+CM | MET/CBT
Number analyzed (Participants) | 51 | 51 | 51
percentage of participants | 58.8 | 64.7 | 35.3

ADVERSE EVENTS:
Arm/Group | MET/CBT+CM/BPT | MET/CBT+CM | MET/CBT
Serious Adverse Events (participants affected / at risk) | 15/51 | 8/51 | 6/51
Other Adverse Events (participants affected / at risk) | 7/51 | 8/51 | 4/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MET/CBT+CM/BPT (N=51) | MET/CBT+CM (N=51) | MET/CBT (N=51)
Residential Treatment for Substance Use (Psychiatric disorders) | 4 (4) | 1 (1) | 2 (2)
Hospitatlization or Residential Treatment for Mental Health (Psychiatric disorders) | 6 (6) | 1 (1) | 1 (1)
Boot Camp, Detention, Incarceration (General disorders) | 4 (4) | 6 (7) | 3 (4)
Overdose (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.96% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MET/CBT+CM/BPT (N=51) | MET/CBT+CM (N=51) | MET/CBT (N=51)
Arrested (General disorders) | 2 (2) | 3 (3) | 1 (1) — Arrest not resulting in boot camp, detention, or incarceration
Running Away (General disorders) | 3 (3) | 2 (2) | 0 (0)
Expelled from School (General disorders) | 2 (2) | 2 (2) | 2 (2)
Dropped Out of School (General disorders) | 0 (0) | 1 (1) | 0 (0)
DCFS Report (General disorders) | 0 (0) | 0 (0) | 1 (1) — Report made to the department of children and family services (DCFS)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No